CLINICAL TRIAL: NCT05736016
Title: Influence of Medial Wedge Corrective Insoles Versus Sham Insoles on Gait Characteristics in Persons After Total Hip Replacement - Randomized Control Trial
Brief Title: Medial Wedge Insoles to Improve Gait in Persons After Total Hip Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STATUT 2020-Reh
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Arthritis of Hip; Fracture of Femur; Aseptic Necrosis; Dysplasia; Hip; Surgical Procedure, Unspecified
Keywords: Total hip replacement; Gait; Insoles; Rehabilitation
MeSH Terms: conditions — Femoral Fractures; Osteonecrosis; Hip Dislocation

STUDY DESIGN:
Intervention Model Description: double-blind sham-controlled single-centre randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants are provided with either active or shame medical devices. Care providers (rehabilitatin team members) and outcome assessors are not acknowledged about patiens' allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Therapy (Active Comparator): Active comparator will undergo a 6-week in-patient rehabilitation aimed at: pharmacologic and non-pharmacologic pain management, improvement of vascular function, cardiopulmonary function, functions of skeletal muscles, range of motion and stability of peripheral joints, gait function, body position, with treadmill walking training being a mandatory part of the program. The rehabilitation program will also address individual needs with psychotherapy and vocational therapy. Follow-up period will be 6 weeks. For the time of the treatment and follow-up period the treatment arm will be provided with individually made corrective medial wedge insoles to be used during all therapeutic and other everyday activities.
  Interventions: Device: medial wedge insoles ((corrective insoles are equipped with hard 10-degree medial wedge, while sham insoles are equipped with pliable 10-degree medial wedge)
- Sham Therapy (Sham Comparator): Sham comparator arm will undergo a 6-week in-patient rehabilitation aimed at: pharmacologic and non-pharmacologic pain management, improvement of vascular function, cardiopulmonary function, functions of skeletal muscles, range of motion and stability of peripheral joints, gait function, body position, with treadmill walking training being a mandatory part of the program . The rehabilitation program will also address individual needs with psychotherapy and vocational therapy. Follow-up period will be 6 weeks. For the treatment and follow-up the control arm will be provided with individually made sham insoles to be used during all therapeutic and other everyday activities.
  Interventions: Device: medial wedge insoles ((corrective insoles are equipped with hard 10-degree medial wedge, while sham insoles are equipped with pliable 10-degree medial wedge)

INTERVENTIONS:
Device: medial wedge insoles ((corrective insoles are equipped with hard 10-degree medial wedge, while sham insoles are equipped with pliable 10-degree medial wedge) — All study participants will be instructed to use insoles for exercising, walking, and other everyday activities.

SUMMARY:
The study will test the hypothesis, that the use of medial wedge insoles in people participating in comprehensive rehabilitation between 1-6 months after total hip replacement, and not having a varus deformity of the knee or symptomatic arthrosis of the medial knee compartment, will improve patient's functioning, the symmetry of gait and stance compared to persons using sham insoles.

The participants will undergo a 6-week program of in-patient rehabilitation aimed at: pharmacologic and non-pharmacologic pain management, improvement of vascular function, cardiopulmonary function, functions of skeletal muscles, range of motion and stability of peripheral joints, gait function, body position. The rehabilitation program will also address individual needs with psychotherapy and vocational therapy.

The study will help to identify correlations between gait parameter change and functional improvement during the rehabilitation following THR.

Study participants will be provided with individually made corrective medial wedge insoles or sham insoles and instructed to use them during gait training and everyday activities.

Functional parameters will be examined at the study entry, at the end of 6 weeks of intervention, and 6 weeks following discharge.

DETAILED DESCRIPTION:
Principal indications for total hip replacement (THR) include hip arthritis - degenerative or inflammatory (91%), fractures of femoral neck (5%), avascular necrosis (2%) and hip dysplasia (2%). Weight-bearing exercises (including treadmill training) are important to improve both impairment and ability to function.

Rationale of testing the effect of medial wedge insoles after THR:

Valgus deformity of the lower limb and insufficiency of the gluteus medius muscle lead to femoral adduction. In patients after a total hip replacement (THR), it will transfer the ground force to the prosthesis cup in the adduction position.

The application of corrective insoles is a simple, inexpensive, and non-invasive intervention that may be easily integrated into daily activities to promote health benefits, provide comfort, and prevent acute and chronic injuries, as well as correct biomechanical deficiencies in the musculoskeletal system (including valgus knee ). An important effect of the insoles is to support the preferred movement pattern and, as a result, reduce unnecessary muscle activity in gait, and decrease fatigue and energy expenditure. The use of insoles can therefore be a valuable addition to gait function exercises. Typically, hindfoot corrective insoles are used with a wedge that corrects the heel between 5-15 degrees. Smaller correction wedge angles are unable to correct the valgus moment and affect the center of pressure (CoP) projection during walking, while wedges with a larger correction angle cause discomfort.[5] Medial wedge insoles increase heel inversion, reduce internal tibial rotation, transfer the CoP medially to the knee joint, and increase the knee and hip abduction moment.

Insufficiency of the gluteus medius muscle causing pelvic descent and internal rotation of the thigh is typical for hip arthritis, especially after THR using the posterior, posterolateral, or direct lateral approach. It was found that the use of medial wedge insoles promotes the activation of the gluteus medius during dynamic activities, although Bird et al. did not confirm this effect in people with low back pain.

Gait symmetry and voluntary walking speed belong to important gait quality parameters measured in patients after THR. Many variables illustrating gait symmetry such as ..step length, step time, time of load changes, foot rotation, time of gait phases, as well as temporal and spatial distribution of forces exerted by specific foot parts may be reliably measured with a treadmill instrumented with force sensors.

To identify publications on the effectiveness of corrective insoles after THR, an analysis of the Pubmed, Medline Central, and Scifinder literature databases was carried out using the key phrase: (("hip" AND ("replace*" OR "plast*" or "simple*")) AND ( "insole*" OR ("foot AND "correc*"))) Identified (November 15, 2019) in databases; Medline Central: 20 records, Scifinder: 73 records, and Pubmed: 66 records. 159 records were reviewed in the title analysis stage, 9 records were eliminated as repeated, 150 records were eliminated as not related to the use of insoles after THR.

Evidence on the usefulness of supination insoles in people with arthritis of the lower limb, and also in people after hip arthroplasty is warranted.

Study design:

A single-center randomized control trial to observe the effect of medial wedge corrective insoles on gait characteristics in persons after THR will be performed in the Rehabilitation Department of the National Institute of Geriatrics, Rheumatology and Rehabilitation, Warsaw, Poland. The trial will involve 100 patients admitted 1-6 months after THR. Consecutive patients fulfilling inclusion criteria will be invited to participate. Participants will be randomly allocated in:

1. Intervention group: the patients will be provided with corrective medial wedge insoles (with hard 10-degree medial wedge)
2. Control group: the patients will be provided with sham medial wedge insoles (with pliable10 degree medial wedge)

Participants' age, sex, time since THR, cause of THR, body height and weight, Q angle, intermalleolar distance, and lower extremities length discrepancy will be measured at the study entry. All insoles will be fabricated individually. The design of insoles will comply with the participant's foot size and needs with regard to lower limb length discrepancy elimination. The participants will be recommended to use the insoles during all therapeutic activities and daily activities during the duration of the program. The participants will undergo a 6-week rehabilitation program provided in the Rehabilitation Department of the National Institute of Geriatrics, Rheumatology and Rehabilitation. The program will be aimed at: pharmacologic and non-pharmacologic pain management, improvement of vascular function, cardiopulmonary function, functions of skeletal muscles, range of motion and stability of peripheral joints, gait function, and body position. The rehabilitation program will also address individual needs with psychotherapy and vocational therapy. The following parameters will be assessed by a blinded researcher in the specific time points (1) 3rd day following delivery of insoles; (2) completion of the 6-week rehabilitation program; (3) follow-up 6 weeks after completion of the rehabilitation program:

Pain intensity (recently and on average during the preceding week), distress produced by pain (recently and on average during the preceding week), and interference of pain with everyday activities (Pain Rating Scale by the British Pain Society, the Polish version; © The British Pain Society 2006), passive ranges of motion of hip, knee, and ankle joints, pain, stiffness, and physical functional disability (Western Ontario and McMaster Universities - WOMAC scale), osteoarthritis-specific symptoms and physical functional disability (The Lequesne OA index), Gait variables: voluntary speed, step time symmetry, time of load change heel to forefoot symmetry, foot rotation symmetry, length symmetry, step width, stance phase symmetry, load response symmetry, single limb support symmetry, swing phase symmetry and variables illustrating the centre of pressure displacement (length of gait line symmetry, single limb support line symmetry, lateral deviation of the center of pressure, anteroposterior position of the center of pressure) (obtained by Zebris Medical Rehawalk software on HP Cosmos Mercury FDM-THP-M2i treadmill), Stance variables: Centre of Pressure path length, 95% confidence ellipse area, symmetry of average forces, Patient's satisfaction with insoles will be assessed at the completion of the study, Dropout rate and adverse effects.

Statistical analysis

Normally distributed data will be described by means and standard deviation and statistically tested using the Student t-test and ANOVA. Data not normally distributed will be described by medians and ranges and statistically tested using non-parametric methods such as Wilcoxon's test and the Kruskal-Wallis test. The frequency will be compared using Fisher's exact test. The normality of data will be tested using the Shapiro-Wilk test. The symmetry of gait and stance will be analyzed using different symmetry indices (such as Symmetry ratio, Symmetry index, Gait asymmetry, and Symmetry angle). The correlations between gait parameter change and functional improvement will be analyzed using Spearman's rank correlations coefficient and Fisher's exact test.

Significance of the results:

The evidence of the beneficial effect of medial wedge insoles on the functioning of patients after THR may result in a recommendation for the use of routine use of such devices after THR. The study will help to identify correlations between gait parameter change and functional improvement during the rehabilitation following THR.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary or secondary hip coxarthrosis or proxmal hip facture
* Total Hip replacement made from posterior or lateral surgical approaches
* Total Hip replacement made less 1-6 months prior to study entry

Exclusion Criteria:

* Total Hip replacement made from anterior or anterolateral approach
* Total Hip replacement made less than 1 month or more than 6 months prior to study entry
* Varus knee (Q angle below 5 degrees in males and below 10 degrees in females
* Symptomatic arthritis of medial compartment of the knee
* Use of corrective insoles (excluding insoles for limb length discrepancy compensation)
* Inability to walk for one minute
* Neurologic conditions
* History of hip prosthesis dislocation
* Cognitive dysfunction (MoCa Score below 26)
* Lack of shoes with a stiff heel counter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in pain according to Pain Rating Scale by the British Pain Society on numeric rating scales at 12 weeks | At baseline and on 12 week
  Pain Rating Scale by the British Pain Society, the Polish version; © The British Pain Society 2006 is a self-reported instrument assessing pain intensity (now and on average last week), distress produced by pain (now and on average last week) and interference of pain with everyday activities. The result is presented on five numeric rating scales ranging from 0 (no pain/distress/interference) to 10 (worst possible pain/distress/interference). Change: (week 12 score - baseline score)
Mean change from baseline in pain, stiffness, and physical functional disability according to Western Ontario and McMaster Universities - WOMAC scale on 12 weeks | At baseline and on 12 week
  WOMAC scale is a self-reported instrument assessing pain, stiffness, and physical functional disability . The results are presented on a numeric scale between 0 (no symptoms, full physical functionning) and 96 (extremely intensive symptoms, extreme disability). Change: (week 12 score - baseline score)
Mean change from baseline in osteoarthritis-specific symptoms and physical functional disability according to Lequesne OA index on 12 weeks | At baseline and on 12 week
  Lequesne OA index is a self-reported instrument assessing osteoarthritis-specific symptoms and physical functional disability. The results are presented on a numeric scale between 0 (no symptoms, full physical functioning) and 24 (extremely intensive symptoms and the worst functioning). Change: (week 12 score - baseline score)

SECONDARY OUTCOMES:
Mean change from baseline in range of motion of lower extremities on 6 weeks | At baseline and on 6 week
  International SFTR Method of Measuring and Recording of Joint Motion (International Standard Orthopaedic Measurements) will be applied to measure the range of motion of the following joints: hip, knee and ankle in operated and non-perated extremity. The results will be provided in degrees. in operated hips flexion above 90 degrees, abduction, internal rotation will not be measured. Normal ranges of motion values are: Hip (nonoperated) S 15 - 0 - 125 (140 degrees); F 45 - 0 - 25 (70 degrees), R 45 - 0 - 40 (95 degrees); Hip (operated): S 15 - 0 - 90 (105 degrees); F 45 - 0 (45 degrees), R 45 - 0 (45 degrees); Knee: S 0 - 0 - 130 (130 degrees); Ankle: S 20 - 0 - 45 (65 degrees) R 20 - 0 - 40 (60 degrees). Change: (week 6 score - baseline score)
Mean change from baseline in range of motion of lower extremities on 12 weeks | At baseline and on 12 week
  International SFTR Method of Measuring and Recording of Joint Motion (International Standard Orthopaedic Measurements) will be applied to measure the range of motion of the following joints: hip, knee and ankle in operated and non-perated extremity. The results will be provided in degrees. in operated hips flexion above 90 degrees, abduction, internal rotation will not be measured. Normal ranges of motion values are: Hip (nonoperated) S 15 - 0 - 125 (140 degrees); F 45 - 0 - 25 (70 degrees), R 45 - 0 - 40 (95 degrees); Hip (operated): S 15 - 0 - 90 (105 degrees); F 45 - 0 (45 degrees), R 45 - 0 (45 degrees); Knee: S 0 - 0 - 130 (130 degrees); Ankle: S 20 - 0 - 45 (65 degrees) R 20 - 0 - 40 (60 degrees). Change: (week 12 score - baseline score)
Mean change from baseline in voluntary gait speed on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure voluntary gait speed. The results can range from 0 to 19,9 km/h. Change (week 6 score - baseline score)
Mean change from baseline in voluntary gait speed on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure voluntary gait speed. The results can range from 0 to 19,9 km/h. Change (week 12 score - baseline score)
Mean change from baseline in step time symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure step time of operated and and non-operated extremity. Symmetry will be calculated as: step time of operated leg/step time of nonperated leg. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in step time symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure step time of operated and and non-operated extremity. Symmetry will be calculated as: step time of operated leg/step time of nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in time of load change heel to forefoot symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure time of load change heel to forefoot. Symmetry will be calculated as: time [sec] of load change heel to forefoot in operated leg/ time of load change heel to forefoot in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in time of load change heel to forefoot symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of load change heel to forefoot. Symmetry will be calculated as: time [sec] of load change heel to forefoot in operated leg/ time of load change heel to forefoot in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in time of maximum force exerted by forefoot symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of maximum force exerted by forefoot. Symmetry will be calculated as: time [sec] of maximum force exerted by forefoot in operated leg/ time of maximum force exerted by forefoot in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in time of maximum force exerted by forefoot symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of maximum force exerted by forefoot. Symmetry will be calculated as: time [sec] of maximum force exerted by forefoot in operated leg/ time of maximum force exerted by forefoot in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in time of maximum force exerted by midfoot symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of maximum force exerted by midfoot. Symmetry will be calculated as: time [sec] of maximum force exerted by midfoot in operated leg/ time of maximum force exerted by midfoot in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in time of maximum force exerted by midfoot symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of maximum force exerted by midfoot. Symmetry will be calculated as: time [sec] of maximum force exerted by midfoot in operated leg/ time of maximum force exerted by midfoot in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in time of maximum force exerted by heel symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of maximum force exerted by heel. Symmetry will be calculated as: time [sec] of maximum force exerted by heel in operated leg/ time of maximum force exerted by heel in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in time of maximum force exerted by heel symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the time of maximum force exerted by heel. Symmetry will be calculated as: time [sec] of maximum force exerted by heel in operated leg/ time of maximum force exerted by heel in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in foot rotation symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the foot rotation. Symmetry will be calculated as: foot rotation [degrees] in operated leg/ foot rotation in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in foot rotation symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the foot rotation. Symmetry will be calculated as: foot rotation [degrees] in operated leg/ foot rotation in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in step length symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the step length. Symmetry will be calculated as: step length [cm] in operated leg/ step length in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in step length symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the step length. Symmetry will be calculated as: step length [cm] in operated leg/ step length in nonperated leg. Possible scores range from 0 to infinity. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in step width on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the step width [cm]. Possible scores range from 0 to 35. Interpretation: interpretation: the lesser step width, the better gait function. Change (week 6 score - baseline score)
Mean change from baseline in step width on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the step width [cm]. Possible scores range from 0 to 35. Interpretation: interpretation: the lesser step width, the better gait function. Change (week 12 score - baseline score)
Mean change from baseline in the length of gait line marked out by the centre of pressure displacement on walking symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the length of gait line marked out by the centre of pressure displacement on walking. Symmetry will be calculated as: length of gait line [mm] in operated leg/length of gait line in nonperated leg. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in the length of gait line marked out by the centre of pressure displacement on walking symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the length of gait line marked out by the centre of pressure displacement on walking. Symmetry will be calculated as: length of gait line [mm] in operated leg/length of gait line in nonperated leg. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in the single limb support line marked out by the centre of pressure displacement on walking symmetry on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the length of the single limb support line marked out by the centre of pressure displacement on walking. Symmetry will be calculated as: single limb support line [mm] in operated leg/ single limb support line in nonperated leg. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in the single limb support line marked out by the centre of pressure displacement on walking symmetry on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the length of the single limb support line marked out by the centre of pressure displacement on walking. Symmetry will be calculated as: single limb support line [mm] in operated leg/ single limb support line in nonperated leg. Possible scores range from 0 to infinity. Perfect symmetry is when the result is 1.0. Higher or lower values reflect asymmetry. Change (week 12 score - baseline score)
Mean change from baseline in lateral deviation of the center of pressure on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the lateral deviation of the center of pressure on walking. Possible scores range from -200 to 200 mm. The lesser lateral deviation, the more symmetrical gait. Change (week 6 score - baseline score)
Mean change from baseline in lateral deviation of the center of pressure on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the lateral deviation of the center of pressure on walking. Possible scores range from -200 to 200 mm. The lesser lateral devaition, the more symmetrical gait. Change (week 12 score - baseline score)
Mean change from baseline in anteroposterior deviation of the center of pressure on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure anteroposterior deviation of the center of pressure (mm). (Possible scores range from -150 to 150. The lesser anteroposterior deviaton, the more balanced gait. Change (week 6 score - baseline score)
Mean change from baseline in anteroposterior deviation of the center of pressure on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure anteroposterior deviation of the center of pressure (mm). (Possible scores range from -150 to 150.The lesser anteroposterior deviaton, the more balanced gait. Change (week 12 score - baseline score)
Mean change from baseline in Centre of Pressure path length in stance on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure Centre of Pressure path length in stance (mm). Possible scores range from 0 to 4800. The shorter path, the more balanced stance. Change (week 6 score - baseline score)
Mean change from baseline in Centre of Pressure path length in stance on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure Centre of Pressure path length in stance (mm). Possible scores range from 0 to 4800. The shorter path, the more balanced stance. Change (week 12 score - baseline score)
Mean change from baseline in 95% confidence ellipse area marked up by the Centre of Pressure displacement in stance on 6 weeks. | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure Centre of Pressure displacement in stance [square mm] Possible scores range from 0 to 125.600. The lesser area, the more stable stance. Change (week 6 score - baseline score)
Mean change from baseline in 95% confidence ellipse area marked up by the Centre of Pressure displacement in stance on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure Centre of Pressure displacement in stance [square mm] Possible scores range from 0 to 125.600. The lesser area, the more stable stance. Change (week 12 score - baseline score)
Mean change from baseline in the ratio of average forces exerted by operated leg in comparison to non-operated leg during stance on 6 weeks | At baseline and on 6 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the he ratio of average forces exerted by operated leg in comparison to non-operated leg during stance. Possible scores range from 0 to 100%. Score 50% - operated leg; 50% non-operated leg reflects symmetrical force distribution. Any deviation reflects stance asymmetry. Change (week 6 score - baseline score)
Mean change from baseline in the ratio of average forces exerted by operated leg in comparison to non-operated leg during stance on 12 weeks | At baseline and on 12 week
  HP Cosmos Mercury FDM-THP-M2i treadmill with Zebris Medical Rehawalk software will be used to measure the he ratio of average forces exerted by operated leg in comparison to non-operated leg during stance. Possible scores range from 0 to 100%. Score 50% - operated leg; 50% non-operated leg reflects symmetrical force distribution. Any deviation reflects stance asymmetry.Change (week 12 score - baseline score)
User's satisfaction with insoles | On 12 week
  (5 point Likert scale will be applied to assess user's satisfaction with insoles the dimension of comfort (how comfortable are the insoles? 2. Very comfortable, 1. Moderately comfortable, 0. Neither comfortable nor uncomfortable, -1. Moderately uncomfortable, -2. Very uncomfortable) and influence on gait (how do insloes influence your gait? 2. Help very much, 1. Help moderately, 0. Neither help nor hamper, -1. Hamper moderately, -2. Hamper very much)
Mean change from baseline in pain according to Pain Rating Scale by the British Pain Society on numeric rating scales at 6 weeks | At baseline and on 6 week
  Pain Rating Scale by the British Pain Society, the Polish version; © The British Pain Society 2006 is a self-reported instrument assessing pain intensity (now and on average last week), distress produced by pain (now and on average last week) and interference of pain with everyday activities. The result is presented on five numeric rating scales ranging from 0 (no pain/distress/interference) to 10 (worst possible pain/distress/interference). Change: (week 6 score - baseline score)
Mean change from baseline in pain, stiffness, and physical functional disability according to Western Ontario and McMaster Universities - WOMAC scale on 6 weeks | At baseline and on 6 week
  WOMAC scale is a self-reported instrument assessing pain, stiffness, and physical functional disability. The results are presented on a numeric scale between 0 (no symptoms, full physical functionning) and 96 (extremely intensive symptoms, extreme disability). Change: (week 6 score - baseline score)
Mean change from baseline in osteoarthritis-specific symptoms and physical functional disability according to Lequesne OA index on 6 weeks | At baseline and on 6 week
  Lequesne OA index is a self-reported instrument assessing osteoarthritis-specific symptoms and physical functional disability. The results are presented on a numeric scale between 0 (no symptoms, full physical functioning) and 24 (extremely intensive symptoms and the worst functioning). Change: (week 6 score - baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Beata Tarnacka, MD PhD, Study Director — National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be made published on Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.

REFERENCES:
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287
- [Background] Robinson RP, Clark JE. Uncemented press-fit total hip arthroplasty using the Identifit custom-molding technique. A prospective minimum 2-year follow-up study. J Arthroplasty. 1996 Apr;11(3):247-54. doi: 10.1016/s0883-5403(96)80074-x. PMID 8713902
- [Background] Mesfin A, Goddard MS, Tuakli-Wosornu YA, Khanuja HS. Total hip and knee arthroplasty in patients with hereditary multiple exostoses. Orthopedics. 2012 Dec;35(12):e1807-10. doi: 10.3928/01477447-20121120-29. PMID 23218641
- [Background] Fukuchi CA, Lewinson RT, Worobets JT, Stefanyshyn DJ. Effects of Lateral and Medial Wedged Insoles on Knee and Ankle Internal Joint Moments During Walking in Healthy Men. J Am Podiatr Med Assoc. 2016 Nov;106(6):411-418. doi: 10.7547/15-077. PMID 28033056
- [Background] Moretti VM, Post ZD. Surgical Approaches for Total Hip Arthroplasty. Indian J Orthop. 2017 Jul-Aug;51(4):368-376. doi: 10.4103/ortho.IJOrtho_317_16. PMID 28790465
- [Background] Hertel J, Sloss BR, Earl JE. Effect of foot orthotics on quadriceps and gluteus medius electromyographic activity during selected exercises. Arch Phys Med Rehabil. 2005 Jan;86(1):26-30. doi: 10.1016/j.apmr.2004.03.029. PMID 15640985
- [Background] Bird AR, Bendrups AP, Payne CB. The effect of foot wedging on electromyographic activity in the erector spinae and gluteus medius muscles during walking. Gait Posture. 2003 Oct;18(2):81-91. doi: 10.1016/s0966-6362(02)00199-6. PMID 14654211
- [Background] Shaw KE, Charlton JM, Perry CKL, de Vries CM, Redekopp MJ, White JA, Hunt MA. The effects of shoe-worn insoles on gait biomechanics in people with knee osteoarthritis: a systematic review and meta-analysis. Br J Sports Med. 2018 Feb;52(4):238-253. doi: 10.1136/bjsports-2016-097108. Epub 2017 Jul 6. PMID 28684391
- [Background] Woodland LH, Francis RS. Parameters and comparisons of the quadriceps angle of college-aged men and women in the supine and standing positions. Am J Sports Med. 1992 Mar-Apr;20(2):208-11. doi: 10.1177/036354659202000220. PMID 1558251
- [Background] Tillman MD, Bauer JA, Cauraugh JH, Trimble MH. Differences in lower extremity alignment between males and females. Potential predisposing factors for knee injury. J Sports Med Phys Fitness. 2005 Sep;45(3):355-9. PMID 16230987
- [Background] Shultz SJ, Nguyen AD, Windley TC, Kulas AS, Botic TL, Beynnon BD. Intratester and intertester reliability of clinical measures of lower extremity anatomic characteristics: implications for multicenter studies. Clin J Sport Med. 2006 Mar;16(2):155-61. doi: 10.1097/00042752-200603000-00012. PMID 16603886
- [Background] Medina McKeon JM, Hertel J. Sex differences and representative values for 6 lower extremity alignment measures. J Athl Train. 2009 May-Jun;44(3):249-55. doi: 10.4085/1062-6050-44.3.249. PMID 19478840
- [Background] Khasawneh RR, Allouh MZ, Abu-El-Rub E. Measurement of the quadriceps (Q) angle with respect to various body parameters in young Arab population. PLoS One. 2019 Jun 13;14(6):e0218387. doi: 10.1371/journal.pone.0218387. eCollection 2019. PMID 31194851
- [Background] Thomas KS, Russell DM, Van Lunen BL, Colberg SR, Morrison S. The impact of speed and time on gait dynamics. Hum Mov Sci. 2017 Aug;54:320-330. doi: 10.1016/j.humov.2017.06.003. Epub 2017 Jun 19. PMID 28641172
- [Background] Fryzowicz A, Dworak LB, Koczewski P. Prophylaxis of medial compartment gonarthrosis in varus knee - current state of knowledge. Arch Med Sci. 2018 Mar;14(2):454-459. doi: 10.5114/aoms.2016.57961. Epub 2016 Mar 29. PMID 29593820
- [Background] Klotzbier TJ, Schott N. Cognitive-Motor Interference during Walking in Older Adults with Probable Mild Cognitive Impairment. Front Aging Neurosci. 2017 Dec 11;9:350. doi: 10.3389/fnagi.2017.00350. eCollection 2017. PMID 29321738
- [Background] Gierus J, Mosiolek A, Koweszko T, Kozyra O, Wnukiewicz P, Loza B, Szulc A. [The Montreal Cognitive Assessment 7.2--Polish adaptation and research on equivalency]. Psychiatr Pol. 2015 Jan-Feb;49(1):171-9. doi: 10.12740/PP/24748. Polish. PMID 25844419
- [Background] Stucki G, Sangha O, Stucki S, Michel BA, Tyndall A, Dick W, Theiler R. Comparison of the WOMAC (Western Ontario and McMaster Universities) osteoarthritis index and a self-report format of the self-administered Lequesne-Algofunctional index in patients with knee and hip osteoarthritis. Osteoarthritis Cartilage. 1998 Mar;6(2):79-86. doi: 10.1053/joca.1997.0097. PMID 9692062
- [Background] Mendiolagoitia L, Rodriguez MA, Crespo I, Del Valle M, Olmedillas H. Kinematic Gait Analysis After Primary Total Hip Replacement: A Systematic Review: Gait After Total Hip Replacement: A Systematic Review. Indian J Orthop. 2020 Apr 16;54(6):767-775. doi: 10.1007/s43465-020-00101-x. eCollection 2020 Nov. PMID 33133399
- [Background] McCrory JL, White SC, Lifeso RM. Vertical ground reaction forces: objective measures of gait following hip arthroplasty. Gait Posture. 2001 Oct;14(2):104-9. doi: 10.1016/s0966-6362(01)00140-0. PMID 11544061
- [Background] Gerhardt JJ, Rondinelli RD. Goniometric techniques for range-of-motion assessment. Phys Med Rehabil Clin N Am. 2001 Aug;12(3):507-27. PMID 11478185
- [Background] Ferguson RJ, Palmer AJ, Taylor A, Porter ML, Malchau H, Glyn-Jones S. Hip replacement. Lancet. 2018 Nov 3;392(10158):1662-1671. doi: 10.1016/S0140-6736(18)31777-X. PMID 30496081
- [Background] Di Monaco M, Castiglioni C. Which type of exercise therapy is effective after hip arthroplasty? A systematic review of randomized controlled trials. Eur J Phys Rehabil Med. 2013 Dec;49(6):893-907, quiz 921-3. Epub 2013 Oct 30. PMID 24172644